CLINICAL TRIAL: NCT06705686
Title: Phase 1 First in Human Trial to Assess Safety and Tolerability of the Novel ACK1 Inhibitor (R)-9b in Patients With Prostate Cancer
Brief Title: Novel ACK1 Inhibitor (R)-9b in Patients With Prostate Cancer
Acronym: PHAROS
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TechnoGenesys, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Washington University School of Medicine (Other); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA286443; 1R01CA286443-01A1 (NIH)
Record Dates: First submitted 2024-11-18; First posted 2024-11-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer (CRPC); Metastatic Castration-resistant Prostate Carcinoma
Keywords: ACK1; TNK2; Non-receptor tyrosine kinase; small molecule inhibitor; prostate cancer; CRPC; kinase inhibitor; Androgen receptor antagonist; Immune modulator
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation: (R)-9bMS (Experimental): Patient will take the assigned dose of (R)-9bMS twice daily by mouth for up to 6 months. Each cycle is 28 days.
  Interventions: Drug: (R)-9bMS
- Expansion: (R)-9bMS (Experimental): Patient will take (R)-9bMS twice daily by mouth for up to 6 months. Each cycle is 28 days. The assigned dose will be determined in the Dose Escalation portion of the trial.
  Interventions: Drug: (R)-9bMS

INTERVENTIONS:
Drug: (R)-9bMS — (R)-9bMS will be given in clinic on day 1, two doses 12 hours (+/- 30 minutes) apart, and on day 2, 12 hours (+/- 30 minutes) after the second day 1 dose. Patients will be admitted overnight for these first 3 doses. Patient must be fasting 1 hour before and 1 hour after doses for these first 3 doses. (R)-9bMS should be taken with a glass of water. Patients will be dispensed home supply after C1D2 morning dose.
  Other Names: Mahatinib

SUMMARY:
TITLE: Phase 1 First in Human Trial to Assess Safety and Tolerability of the Novel ACK1 Inhibitor (R)-9bMS in Patients with Prostate Cancer (PHAROS)

STUDY DESCRIPTION: Prostate cancer (PC) patients receive androgen deprivation therapy (ADT), but recalcitrant disease recurs typically within 2-3 years, referred to as the Castration Resistant Prostate Cancer (CRPC). Androgen receptor (AR) targeted therapies, such as Enzalutamide (Enz) or Abiraterone (Abi), are FDA-approved therapeutics for CRPC patients. However, virtually all patients develop resistance.

A non-receptor tyrosine kinase, ACK1 act as a novel epigenetic modifier in prostate tumors, regulating AR and its splice variant, AR-V7 expression. A new class of ACK1 small molecule inhibitor, (R)-9bMS, was developed that exhibited excellent drug-like properties. Treatment with (R)-9bMS suppressed Abi and Enz-resistant tumor growth in mice. Robust immune activation against prostate tumors was also reflected in mice treated with ACK1 inhibitor, (R)-9bMS. Importantly (R)-9bMS functionally reinvigorated peripheral blood mononuclear cells (PBMCs) of CRPC patients to mount a robust immune response against CRPC organoids. Collectively, these data indicate that the ACK1 inhibitor, (R)-9bMS, fulfills a unique niche, wherein it not only suppressed AR/AR-V7 within the tumor milieu, but also activated host immune system by overcoming CSK-restrained LCK activity, to mount a robust 'dual' anti-tumor response.

OBJECTIVES: Primary Objective: To assess the safety and tolerability of (R)-9bMS in patients with metastatic castration-resistant prostate cancer.

Secondary Objectives: To determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of (R)-9bMS in patients with CRPC. To determine the pharmacokinetics (PK) of (R)-9bMS in patients after single and multiple dose oral administration. To assess clinical outcomes and anti-tumor activity in patients treated with (R)-9bMS.

ENDPOINTS: Primary Endpoint: Frequency of dose-limiting toxicities and toxicity and severe AEs per CTCAE v 5.0.

Secondary Endpoints:

* RP2D (recommended phase 2 dose)
* PK (pharmacokinetics)
* PSA responses
* Duration of responses
* ORR (objective response rate)
* OS (overall survival)
* PFS (progression free survival)
* DSS (disease specific survival)
* Toxicity and severe AEs per CTCAE v 5.0 STUDY POPULATION: Approximately 18-30 adult patients with a histologic or cytologic diagnosis of metastatic castration resistant prostate cancer will be enrolled.

PHASE: Phase I

DESCRIPTION OF SITES: This study will be open to enrollment at the University of Wisconsin Carbone Cancer Center

DESCRIPTION OF STUDY INERVENTION: (R)-9bMS will be taken by mouth twice daily until completion of 12 cycles, progression or intolerance

STUDY DURATION: 12 months for enrollment + 12 months treatment + 12 months follow-up + 12 months for data analysis = 48 months.

DETAILED DESCRIPTION:
ACK1/TNK2, a non-receptor tyrosine kinase contributes to prostate cancer pathophysiology. Activated ACK1 expression is significantly correlated with the severity of disease progression. In spite of the considerable clinical significance of pathogenic ACK1 activation in prostate [and lung & breast] cancers, no ACK1 inhibitor has been tested in clinical trials to date. ACK1 inhibitor, (R)-9bMS, also known as (R)-9b, with IC50 of 13 nM, suppresses AR/AR-V7 levels and sensitizes Enz-resistant CRPCs.

STUDY DESIGN: This phase Ib single-center open-label The PHAROS trial, "Phase 1 First in Human Trial to Assess Safety and Tolerability of the Novel ACK1 Inhibitor (R)-9bMS in Patients with Prostate Cancer", will establish the safety/tolerability and recommended phase II dosing (RP2D) for (R)-9bMS. Given the unique cancer suppressing properties of the (R)-9bMS compound, its safety and tolerability and proposed Phase 2 dosing will be evaluated in a first-in-human trial in CRPC patients who have stopped responding to Enz or Abi. Post-treatment PSA levels and radiographic responses will be assessed, which will provide preliminary assessment of the efficacy; immune responses will be evaluated, which will provide exploratory assessment immunomodulation.

JUSTIFICATION FOR DOSE: (R)-9bMS will be administered orally twice a day, with an interval of 12 hours between doses.

Both the 28-day rat and 28-day dog toxicity studies were conducted using the clinically-relevant mesylate salt (MS) form of the (R)-9b drug substance.

The results of the 28-day definitive toxicity studies were used to calculate a reasonably safe clinical starting dose for (R)-9bMS in the planned Phase 1 trial. The approach used is consistent with guidance provided in the ICH S9 guideline and the Senderowicz 2010 publication and involves setting the starting dose at 1/10th of the STD10 in rodents. If the nonrodent is the most appropriate species, then 1/6th of the HNSTD is considered an appropriate starting dose.

Step #1: Identifying the rodent STD10 and nonrodent HNSTD values In the 28-day toxicity studies conducted in rats and dogs, the STD10 and HNSTD values were identified as 60 mg/kg/day (R)-9bMS and 45 mg/kg/day (R)-9b, respectively.

* Rat STD10 = 60 mg/kg/day (R)-9bMS
* Dog HNSTD = 33.3 mg/kg/day (R)-9b [41.3 mg/kg/day (R)-9bMS]

Step #2: Converting the STD10 and HNSTD dosages from units of mg/kg/day to units of mg/m2/day:

* Rat STD10 = 60 mg/kg/day X 6 (rat km value) = 360 mg/m2/day (R)-9bMS
* Dog HNSTD = 33.3 mg/kg/day X 20 (dog km value) = 666 mg/m2/day (R)-9b [825.8 mg/kg/day (R)-9bMS]

Step #3: The safe starting dose in humans is 1/10th of the rat STD10 or 1/6th of the dog HNSTD:

* Rat STD10 = 360 mg/m2/day ÷ 10 = 36.0 mg/m2/day (R)-9bMS
* Dog HNSTD = 666 mg/m2/day ÷ 6 = 111 mg/m2/day (R)-9b [137.6 mg/kg/day (R)-9bMS]

Step #4: The lower of the two dosages (in mg/m2/day) is identified as the starting dose in humans:

• 36.0 mg/m2/day < 111 mg/m2/day

For an average 60-kg individual with a body surface area of 1.62 m2, this would be a daily dose of 58.32 mg (R)-9bMS (36.0 mg/m2/day X 1.62 m2).

One capsule containing 30 mg will be administered twice a day to patients for a total daily dose of 60 mg for the level 1 dose.

The phase I trial adopts a Bayesian optimal interval (BOIN) design for dose escalation/stay/de-escalation. If excessive dose limiting toxicities are observed at the first dose level requiring dose reduction, the (R)-9bMS dose will be reduced to 30 mg/day. If no excessive toxicities are observed, the dose will escalate gradually following the decision rules dictated to 300 mg/day in five phases. The trial expects a maximum of 40 patients.

STRATEGIES FOR RECRUITMENT AND RETENTION Subjects seen in the Medical Oncology clinics of the UWCCC with metastatic, castration-resistant prostate cancer, previously treated with 2nd generation AR targeted therapies, who have disease progression who meet the eligibility criteria will be recruited. A detailed explanation of the risks and benefits of the study will be provided, and informed consent will be obtained. Follow up will be performed as detailed below to ensure close monitoring of safety and for evidence of side effects.

TREATMENT PLAN Plan of Treatment: For chemistry panel, the following labs will be performed: Albumin, ALP, amylase, ALT, AST, bicarbonate, BUN, chloride, creatinine, glucose, calcium, LDH, lipase, magnesium, phosphorus, potassium, sodium, total bilirubin, and total protein.

For hematology panel, the following labs will be performed: WBC count w/differential (neutrophils, basophils, eosinophils, lymphocytes, monocytes), hematocrit, platelet count, RBC count, hemoglobin Symptoms assessment involves review of systems for adverse effects monitoring and toxicity grading as per NCI Common Terminology Criteria for Adverse Events (v. 5). Screening (performed within 28 days of Day 1 unless otherwise noted)

1. Confirm potential eligibility by history, pathology, diagnosis, and serum PSA levels
2. CT scan of chest, abdomen and pelvis; bone scan
3. Sign consent form
4. Physical examination, including vital signs, symptoms assessment, and ECOG performance score
5. 12-lead ECG
6. Hematology and chemistry panels and serum testosterone
7. Serum PSA
8. 100 ml peripheral blood (green-top heparinized tubes) for research
9. Biopsy of metastatic site for research (only for patients treated in MTD expansion cohort)

END OF TREATMENT (EOT)

1. Physical examination, including vital signs, weight, adverse event assessment, concomitant medications, and ECOG performance score
2. Blood draw for hematology and chemistry panels, testosterone and PSA
3. 12-lead ECG
4. 100 mL peripheral blood (green-top heparinized tubes) for research

DOSE ESCALATION SCHEMA Level -1 30 mg PO QD; total 30 mg daily (1 capsule per day) Level 1 (Starting Dose) 30 mg PO BID; total 60 mg daily (2 capsules per day) Level 2 60 mg PO BID; total 120 mg daily (4 capsules per day) Level 3 90 mg PO BID; total 180 mg daily (6 capsules per day) Level 4 120 mg PO BID; total 240 mg daily (8 capsules per day) Level 5 150 mg PO BID; total 300 mg daily (10 capsules per day)

DEFINITION OF MTD, DLT and DOSE ESCALATION CRITERIA The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which two patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity during the first cycle. Dose escalations will proceed until the MTD has been reached.

Dose Limiting Toxicities (DLTs)

* DLTs are defined as any (R)-9bMS related (TRAE) toxicity that are ≥ Grade 3 occurring within the 28 days post (R)-9bMS treatment (starting with first day of dosing), with the following caveats:
* Any ≥ Grade 3 hematologic toxicities EXCEPT:

  * Grade 3 neutropenia lasting < 7 days
  * Grade 3 thrombocytopenia without bleeding or requiring platelet transfusion
* Any ≥ Grade 3 Non-hematologic toxicities EXCEPT:

  * Grade 3 nausea, vomiting and/or diarrhea lasting < 72 hours
  * Grade 3 fatigue lasting < 7 days
  * Any non-hematologic Grade 3 clinical laboratory AE that is asymptomatic and returns to ≤ Grade 2 within 72 hours * Asymptomatic Grade 3 electrolyte abnormalities, symptomatic Grade 3 abnormalities that persist >72 hours despite appropriate replacement therapy will be considered a DLT
* Additionally, the following events will be considered DLTs if they occur during the first cycle:

  * Any Grade 5 toxicity
  * Any death not clearly due to the underlying disease or extraneous causes
  * Any event that meets Hy's law criteria
  * Delay in Cycle 2 due to toxicity by > 14 days

DURATION OF THERAPY

In the absence of treatment delays due to adverse events, treatment may continue for up to 1 year or until one of the following criteria applies:

* Documented and confirmed disease progression
* Death
* Adverse event(s) that, in the judgment of the investigator, may cause severe or permanent harm or which rule out continuation of study drug
* Specific conditions described in the dose modifications section
* If the subject does not recover from his toxicities to tolerable grade ≤ 2 within 6 weeks, the subject will have study treatment discontinued
* Inability to tolerate the minimum protocol-specified dose of study treatment
* Participation in another clinical study using an investigational agent, investigational medical device, or other intervention
* General or specific changes in the patient's condition render the patient unable to receive further treatment in the judgment of the investigator
* Serious noncompliance with the study protocol
* Patient withdraws consent
* Request by regulatory agencies for termination of an individual subject or all subjects under the protocol

DURATION OF FOLLOW-UP Patients will have a safety follow-up visit or a review of the medical record at 12 months to assess disease and survival status.

DATA AND SAFETY MONITORING PLAN

The entities providing oversight of safety and compliance with the protocol require reporting, as outlined below. Adverse events (AE) include the following:

1. An exacerbation, or an unexpected increase in frequency or intensity of a pre-existing condition, including intermittent or episodic conditions.
2. Significant or unexpected worsening or exacerbation of the condition/indication under investigation.
3. A suspected drug interaction.
4. An intercurrent illness.
5. Any clinically significant laboratory abnormality.

Serious adverse events (SAE) are any events occurring that result in any of the following outcomes:

1. Subject death
2. Life-threatening adverse event
3. Inpatient hospitalization or prolongation of existing hospitalization
4. Persistent or significant disability/incapacity
5. Congenital anomaly or birth defect

A life-threatening event is defined as any adverse event that places the subject, in the view of the investigator, at immediate risk of death from the reaction.

* Is another important medical event
* Is a new cancer
* Is associated with an overdose.

SEVERITY RATING/GRADING SCALE: Adverse events are classified by organ system and graded by severity according to the current NIH Common Terminology Criteria V. 5. The defined grades use the following general guidelines:

* 0 No adverse event or within normal limits
* 1 Mild adverse event
* 2 Moderate adverse event
* 3 Severe adverse event
* 4 Life-threatening or disabling adverse event
* 5 Fatal adverse event

All adverse events will be recorded from time of treatment initiation through 30 days after the final dose of study treatment, as well as any time after these 30 days for events that are believed to be at least possibly related to study treatment.

B. Disease Oriented Team Meetings UWCCC site: This study undergoes review of subject safety at regularly scheduled Disease Oriented Team (DOT) meetings where the following are discussed as applicable: number of subjects enrolled, subject treatments given, dose holds/modifications, significant toxicities, response to treatment, and the subjects' overall status. These discussions are documented in the DOT meeting minutes.

C. UWCCC Data and Safety Monitoring Committee (DSMC) Study Progress Review and Oversight The review of Protocol Summary Reports (PSRs) enables the UWCCC DSMC to assess whether the study should continue, continue with modifications, be suspended, or be closed. Following their review, the UWCCC DSMC will notify the sponsor-investigator of their recommendation and the authority for continuing, modifying, suspending, or closing the protocol is the responsibility of the applicable sponsor-investigator, Principal Investigator, IRB, FDA or other regulatory authority associated with the protocol.

Based on the risk level of this study, as determined by the UWCCC Protocol Review and Monitoring Committee, PSRs must be submitted to the UWCCC DSMC by the UWCCC site on a quarterly basis.

The UWCCC site is responsible for ensuring participating sites enter data used to populate the PSRs in a timely manner into the UWCCC instance of OnCore. These data include: accrual information, Serious Adverse Events (SAEs), response to treatment, events reportable to IRB (e.g., non-compliance, unanticipated problems).

1. UWCCC DSMC Review of Auditing and/or Monitoring Reports Reports created through the auditing and/or monitoring activities at all sites are submitted in real-time by the UWCCC site to the UWCCC DSMC. Summary data and/or query reports are submitted in lieu of detailed reports. Following the review of these reports, the committee may issue a request for corrective and/or preventive action(s), protocol suspension, or for-cause audit(s).
2. UWCCC DSMC Review of Non-compliance, Unanticipated Problems, and Other IRB Reportable Events UWCCC site: Reports of non-compliance, unanticipated problems, and other IRB reportable events are submitted to the IRB of record for the study and to the UWCCC DSMC, via an email to DSMC@carbone.wisc.edu, simultaneously.
3. Real-time UWCCC DSMC Review of Serious Adverse Events (SAEs) The UWCCC DSMC Chair, or designee, reviews all SAEs occurring on the study, regardless of site, to determine if immediate action is required.

UWCCC site: The Principal Investigator (PI), or designee, notifies the following individuals/entities of SAEs as applicable:

* Other investigators involved with the study at the UWCCC
* IRB of record for the study conducted at the UWCCC, per the IRB's reporting requirements
* UWCCC DSMC
* Medical Monitor: Dr. Saurabh Rajguru
* Sponsor (TechnoGenesys): Dr. Gerald Andriole o Email: jerry@technogenesys.com

D. Serious Adverse Event Reporting Serious Adverse Events Requiring 24-Hour Reporting UWCCC site: All Serious Adverse Events must be reported within 24 hours to the UWCCC DSMC Chair via an email to saenotify@uwcarbone.wisc.edu within one business day. The OnCore SAE Details Report must be submitted along with other report materials as appropriate (FDA Medwatch Form #3500, UWCCC routing form, de-identified supporting documentation available at that time of initial reporting).

E. Sponsor Responsibilities for SAE Review

The sponsor (i.e., TechnoGenesys IND holder) will have the responsibilities of the study sponsor in accordance with FDA 21 CFR 312.32. In this capacity, the sponsor reviews all reports of serious adverse events occurring on the study and makes a documented determination of 1) suspectedness (i.e., whether there is a reasonable possibility that the drug caused the AE); and 2) unexpectedness (the event is not listed in the Investigator's Brochure or is not listed at the specificity or severity that has been observed) in the context of this study. SAE with suspected causality to study drug and deemed unexpected are reported as IND Safety Reports by the sponsor, or designee, to the following within 15 calendar days unless otherwise designated below:

* FDA
* All participating investigators on the study, and the external global sponsor (if applicable).
* Other oversight committees (NIH OSP) All fatal or life-threatening SAE that are unexpected and have suspected causality to the study drug will be reported by the Sponsor (TechnoGenesys), or designee, to the following within 7 calendar days: Dr. Gerald Andriole; Email: jerry@technogenesys.com

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed prostate cancer (mCRPC).
2. Must have evidence of metastatic disease on conventional imaging (eg. CT, MRI, technetium bone scan). May have any type or location of metastases (bone, lymph node, visceral). RECIST 1.1 measurable disease is not required; may have bone-only metastases.
3. Ongoing androgen deprivation therapy (ADT) at time of study enrollment (GnRHR agonist such as leuprolide, goserelin, triptorelin, buserelin, histrelin; GnRHR antagonists such as degarelix or relugolix), or history of surgical castration.
4. Must have evidence of castrate testosterone levels with baseline serum testosterone level of 50 ng/dL or less at time of study start, and castrate levels should be maintained throughout study.
5. Evidence of progressive castration-resistant prostate cancer, defined as at least 2 consecutive rises of PSA, at least 1 week apart with the last PSA ≥ 2 ng/mL or by evidence of radiographic progression.
6. Patients must have had prior disease progression on at least one novel hormonal agent (NHA) (eg enzalutamide, abiraterone, apalutamide, darolutamide, etc.); treatment with NHA could have occurred in the castration-sensitive or castration-resistant setting.
7. Prior palliative radiation therapy for bone metastasis (must be complete ≥ 14 days prior to enrollment) or any other radiation therapy (must be complete ≥ 28 days prior to enrollment) is allowed. Prior definitive radiation therapy for localized prostate cancer is allowed.
8. Recovery to baseline or ≤ grade 1 from toxicities related to any prior treatments, unless AEs are clinically nonsignificant and/or stable on supportive therapy.
9. At least 18 years of age.
10. ECOG performance status ≤ 1
11. Normal bone marrow and organ function as defined below:

    * Absolute neutrophil count ≥ 1,500/mm3 without granulocyte colony-stimulating factor support
    * White blood cell count ≥ 2,000/mm3
    * Platelets ≥ 100,000/mm3 without transfusion
    * Hemoglobin ≥ 9.0 g/DL
    * Total bilirubin ≤ 1.5 x IULN (for subjects with Gilbert's disease ≤ 3.0 x IULN)
    * AST(SGOT), ALT(SGPT) ≤ 3.0 x IULN
    * Serum creatinine ≤ 1.5 x IULN or calculated creatinine clearance ≥ 45 mL/min by Cockcroft-Gault
    * Serum albumin ≥ 2.8 g/dL
    * Urine protein/creatinine ration (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol) (only evaluated if creatinine abnormal per criteria above
    * PT/INR or PTT < 1.5 x IULN (PT/INR must be drawn < 7 days prior to biopsy for those patients treated in MTD cohort), unless participant is receiving anticoagulant therapy and these are within intended therapeutic ranges for anticoagulant.
12. Corrected QT interval calculated by the Fridericia formula (QTcF) ≤ 500 ms (by ECG).
13. Ability to understand and willingness to sign an IRB approved written informed consent document (or that of the legally authorized representative, if applicable).
14. Willingness and ability to undergo biopsy for research component of the trial (for patients treated in MTD cohort)
15. Heterosexually active male patients (along with their female partners) are required to use two forms of acceptable contraception, including one barrier method, during participation in the study and for 5 months following the last day of study treatment. If a female partner of a male patient becomes pregnant during therapy or within 5 months after the last day of study treatment, the investigator must be notified in order to facilitate outcome follow-up.

Exclusion Criteria:

1. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 14 days before first dose of study treatment.
2. Exclusively small cell variant of prostate cancer, or other prostate cancer histology that does not contain adenocarcinoma
3. Inability to swallow pills.
4. Presence of a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 calendar days of start of study treatment. Inhaled or topical steroids and adrenal replacement steroid doses < 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
5. Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to first dose of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, or superficial bladder cancer. Any history of prior malignancy must be reviewed by the PI.
6. Currently receiving any other investigational agents.
7. Any anti-androgen receptor agents or abiraterone (or similar CYP17,20 lyase inhibitor) within 14 days or 5 half-lives, whichever is longer, prior to the start of study drug.
8. Use of Radium-223 or other radioligand/radiopharmaceutical within 28 days prior to the start of study drug
9. Any gastrointestinal issues affecting absorption (e.g. gastrectomy, bowel resection, etc), as determined by the PI.
10. Blood transfusion within 28 days of screening.
11. Use of hormonal agents or supplements with potential anti-tumor activity against prostate cancer, as determined by the PI, within 28 days prior to the start of study drug.
12. Bone-modifying agents (eg zolendronic acid, denosumab, etc) may not be initiated after start of study drug; previously initiated agents may be continued while on trial.
13. Patients with known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks prior to first dose of study treatment after radiotherapy or at least 4 weeks prior to first dose of study treatment after major surgery (e.g., removal or biopsy of brain metastasis). Eligible subjects must be neurologically asymptomatic.
14. History of seizures or seizure disorder.
15. A history of allergic reactions attributed to compounds of similar chemical or biologic composition to (R)-9bMS used in the study.
16. Uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

    * Cardiovascular disorders:

      * Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
      * Uncontrolled hypertension defined as sustained blood pressure (BP) > 160 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.
      * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic events, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within six months before the first dose of study treatment.

        * Subjects with a diagnosis of incidental, subsegmental PE or DVT within six months are allowed if stable, asymptomatic, and treated with anticoagulation for at least 1 week before the first dose of study treatment.
    * Gastrointestinal (GI) disorders associated with a high risk of perforation or fistula formation, as determined by the PI:

      * The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.
      * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within six months before the first dose.

    Note: Complete healing of an intra-abdominal abscess must be confirmed before the first dose.
    * Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before the first dose.
    * Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
    * Lesions invading or encasing any major blood vessels.
    * Other clinically significant disorders that would preclude safe study participation.

      * Serious non-healing wound/ulcer/bone fracture.
      * Uncompensated/symptomatic hypothyroidism.
      * Moderate to severe hepatic impairment (Child-Pugh B or C).
17. Active hepatitis B or C or active HIV per review of medical records. Patients with well-controlled HIV or hepatitis B or C, or who have had curative treatment for hepatitis C, may be considered if they meet all other criteria and after discussion with the PI using the following criteria for guidance:

    https://www.fda.gov/media/121319/download
18. History of organ allograft.
19. Major surgery (e.g., GI surgery removal or biopsy of brain metastasis) within eight weeks before the first dose of study treatment. Complete wound healing from major surgery must have occurred one month before the first dose and from minor surgery (e.g., simple excision, tooth extraction) at least ten days before the first dose (with the exception of the baseline biopsy, which must have occurred no less than 6 days prior to the first dose). Patients with clinically relevant ongoing complications from prior surgery are not eligible.
20. Any other medical intervention or condition, which, in the opinion of the PI or treating physician, could compromise patient safety or adherence with the study requirements (including biopsies), or confound results of the study, over the treatment period.
21. Any known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
22. Patients cannot have concurrent enrollment on other phase I, II, or III investigational treatment studies in which they are actively receiving treatment (participation in long-term follow-up is acceptable).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of dose-limiting toxicities (Dose Escalation only) | From day 1 of treatment through day 28 of treatment
  Dose-limiting toxicities are defined in the protocol.

SECONDARY OUTCOMES:
Recommended phase 2 dose (RP2D) (Dose Escalation only) | From day 1 of treatment through day 28 of treatment
  RP2D has traditionally been synonymous with the highest safe dose, or maximum tolerated dose (MTD) as determined based on, but can be lower than MTD based on comprehensive review of all available data from the phase I study (including dose limiting toxicity data, pharmacodynamic (PD)/pharmacokinetic (PK) study and efficacy data).
Number of patients with a prostate specific antigen (PSA) response | From baseline through end of treatment (up to 6 months)
  PSA response is defined by at least 50% decline in PSA level from baseline measured twice at least 3 weeks apart.
Overall response rate (ORR) | From baseline through end of treatment (up to 12 months)
  ORR is defined as proportion of patients achieving complete response (CR) and partial response (PR) by RECIST 1.1 or by PCWG3 criteria.
Progression-free survival (PFS) | From start of treatment through the completion of follow-up (up to 24 months)
  PFS is defined from date of first treatment to date of progression or death or last follow-up, whichever is earlier.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas McNeel, MD, PhD, Study Director — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center (UWCCC) - Cancer Connect, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sawant M, Mahajan K, Renganathan A, Weimholt C, Luo J, Kukshal V, Jez JM, Jeon MS, Zhang B, Li T, Fang B, Luo Y, Lawrence NJ, Lawrence HR, Feng FY, Mahajan NP. Chronologically modified androgen receptor in recurrent castration-resistant prostate cancer and its therapeutic targeting. Sci Transl Med. 2022 Jun 15;14(649):eabg4132. doi: 10.1126/scitranslmed.abg4132. Epub 2022 Jun 15. PMID 35704598
- [Background] Chouhan S, Sawant M, Weimholt C, Luo J, Sprung RW, Terrado M, Mueller DM, Earp HS, Mahajan NP. TNK2/ACK1-mediated phosphorylation of ATP5F1A (ATP synthase F1 subunit alpha) selectively augments survival of prostate cancer while engendering mitochondrial vulnerability. Autophagy. 2023 Mar;19(3):1000-1025. doi: 10.1080/15548627.2022.2103961. Epub 2022 Jul 27. PMID 35895804
- [Background] Sridaran D, Chouhan S, Mahajan K, Renganathan A, Weimholt C, Bhagwat S, Reimers M, Kim EH, Thakur MK, Saeed MA, Pachynski RK, Seeliger MA, Miller WT, Feng FY, Mahajan NP. Inhibiting ACK1-mediated phosphorylation of C-terminal Src kinase counteracts prostate cancer immune checkpoint blockade resistance. Nat Commun. 2022 Nov 14;13(1):6929. doi: 10.1038/s41467-022-34724-5. PMID 36376335
- [Background] Mahajan NP, Coppola D, Kim J, Lawrence HR, Lawrence NJ, Mahajan K. Blockade of ACK1/TNK2 To Squelch the Survival of Prostate Cancer Stem-like Cells. Sci Rep. 2018 Jan 31;8(1):1954. doi: 10.1038/s41598-018-20172-z. PMID 29386546
- [Background] Mahajan K, Malla P, Lawrence HR, Chen Z, Kumar-Sinha C, Malik R, Shukla S, Kim J, Coppola D, Lawrence NJ, Mahajan NP. ACK1/TNK2 Regulates Histone H4 Tyr88-phosphorylation and AR Gene Expression in Castration-Resistant Prostate Cancer. Cancer Cell. 2017 Jun 12;31(6):790-803.e8. doi: 10.1016/j.ccell.2017.05.003. PMID 28609657